CLINICAL TRIAL: NCT05120245
Title: Fertility Preservation in Transgender Persons: a Retrospective Look At the Decision and a Survey of the Desire for Children.
Brief Title: Fertility Preservation in Transgender Persons: a Retrospective Look
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: BC-09136
Record Dates: First submitted 2021-09-15; First posted 2021-11-15 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Fertility Preservation in Transgender Persons

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Patients in this study will be asked how they feel about the decision to freeze gametes, using a validated questionnaire. In addition, a number of questions with free text fields will be included in the questionnaire to write down any reasons for their satisfaction or regret. In a second part, the intention to use the frozen material will be assessed. We focus on techniques with real perspectives (e.g. cryopreservation of oocytes and sperm cells) and not on techniques that are more experimental for later use (cryopreservation of ovarian and testicular tissue).

ELIGIBILITY:
Inclusion Criteria:

* Dutch speaking
* Sperm or oocyte preservation between june 2015 and june 2020. Survey in 2021

Exclusion Criteria:

* Ovarian and testicular tissue cryopreservation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: transgender personen
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Transgender people's retrospective view of the decision | fertility preservation between june 2015 and june 2020 (5 years). Survey in 2021 (up to 7 years after preservation)
  Study of transgender persons' retrospective evaluation of the decision to freeze egg or sperm cells prior to gender-confirming hormonal or surgical treatment in transition
Satisfaction/ regret about the decision | fertility preservation between june 2015 and june 2020 (5 years). Survey in 2021 (up to 7 years after preservation)
  Survey on the reasons for satisfaction/ regret regarding the decision to freeze egg cells or sperm cells prior to gender-confirming hormonal or surgical treatment in the context of transition
Intention | fertility preservation between june 2015 and june 2020 (5 years). Survey in 2021 (up to 7 years after preservation)
  Examination of the intention to use the frozen egg cells or sperm cells to fulfil a desire to have children

CONTACTS AND LOCATIONS:
Overall Officials: Stoop, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No